CLINICAL TRIAL: NCT03493347
Title: A Mixed Methods Investigation of Equine-assisted Occupational Therapy for Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Wendy Wood, Director of Research, Temple Grandin Equine Center, Colorado State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-7112H
Record Dates: First submitted 2018-03-26; First posted 2018-04-10 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: multiple baseline single case experimental design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Equine-assisted Occupational Therapy (Experimental): All children will receive the Equine-assisted Occupational Therapy (EAOT) intervention, which includes occupational therapy administered in an equine environment. Common intervention activities include grooming, tacking, mounting, and riding the horse.
  Interventions: Behavioral: Equine-assisted Occupational Therapy

INTERVENTIONS:
Behavioral: Equine-assisted Occupational Therapy — Occupational therapy provided in an equine environment that includes activities such as groundwork, grooming, tacking, mounting, and riding horses

SUMMARY:
Children with autism spectrum disorders (ASD) often participate in equine-assisted interventions, where practitioners partner with horses to improve the health and well-being of the clients they serve. One of these interventions is equine-assisted occupational therapy (EAOT). The first aim of this study is to assess the effectiveness of EAOT at improving the social, behavioral, and occupational functioning of children with ASD. Second, this study aims to conceptually develop the theory of change that guides how horses are integrated into occupational therapy for children with ASD. Eight children with ASD will participate in 10 weeks of EAOT. The quantitative strand will involve caregivers filling out measures of social functioning, self-regulation, and occupational performance on a weekly basis. Investigators hypothesize children will demonstrate improved performance on these measures during the intervention in comparison to baseline. The qualitative strand will consist of interviews with the providing occupational therapists aimed at understanding the theory behind why the intervention is effective. The results of this study will have implications for children with ASD, their families, and occupational therapists providing services to individuals with ASD.

DETAILED DESCRIPTION:
The proposed study will implement a mixed-methods investigation of equine-assisted occupational therapy (EAOT) for children with autism spectrum disorder (ASD).

QUANTIATIVE STRAND

PARTICIPANTS Investigators will distribute fliers to local schools and ASD organizations to recruit eight participants for the study. Investigators will screen children for inclusion through a four-step process. They will call interested participants to ensure eligibility for the study, provide basic information, and answer any questions. Next, investigators will mail interested participants a packet that includes the SCQ, the ABC-C, and Hearts and Horses Enrollment Packet, along with a cover letter and instructions to mail back the completed forms, which will include a physician's signature stating the child is medically cleared to ride horses. Next, eligible participants will attend a screening at Hearts and Horses Therapeutic Riding Center to ensure they meet all PATH, Intl standards, and can ride a horse for 10 minutes while following safety rules. Finally, eligible participants will attend a final screening visit that will include administration of the ADOS-2, Leiter-3, and Adaptive Behavior Assessment System, Third Edition (ABAS-3). Eight participants who meet criteria will be enrolled.

SCREENING MEASURES. Social Communication Questionnaire (SCQ). This parent-report measure is a quick, 10-minute screen for ASD. A score of 15 or above indicates the individual likely has ASD. The SCQ has strong discrimination between children with and without ASD and is widely used for entry into ASD research studies.

Autism Diagnostic Observation Schedule, Second Edition (ADOS-2). The ADOS- 2 is a play-based assessment of communication, social interaction and behaviors, and is often used to confirm a clinical diagnosis of ASD. The ADOS has strong predictive validity for diagnosis of ASD. Participants who meet clinical-cutoffs for ASD will be included in the study. The ADOS-2 requires extensive training to administer reliably; an investigator who has obtained research-level reliability will administer the ADOS-2 to potential participants.

Leiter International Performance Scales, Third Edition (Leiter-3). The Leiter-3 is a completely nonverbal measure of intelligence and cognitive abilities that is widely used with the ASD population. The Brief IQ score can be used reliably in place of the Full IQ score when a minimal IQ estimate is needed; therefore, this study will use the Brief IQ version of the Leiter-3. Participants who have an IQ below 55 will be excluded from the study. A registered and licensed occupational therapist will administer the Leiter-3.

Aberrant Behavior Checklist- Community (ABC-C). The ABC-C is a valid and reliable behavior rating scale that measures the extent of problem behaviors in children and adults with development disabilities. Any adult who knows the child well, in this case the caregiver, can complete the 58-item checklist. The irritability and hyperactivity subscales will be used as outcome measures in the study. Therefore, to avoid a ceiling effect as described above, children included in this study must have a combined score ≥ 11 on the irritability and hyperactivity subscales of the ABC-C, as established by Gabriels et al. (2015).

PATH, Intl. Standards. PATH, Intl provides a list of contraindications for participants who should not participate in equine-assisted interventions. In order to ensure participants meet all PATH, Intl standards, they will complete Hearts and Horses enrollment packet and process.

Adaptive Behavior Assessment System (ABAS-3). The ABAS-3 is a norm-referenced rating scale that measures ten domains of adaptive behaviors and can be completed by a caregiver. The ABAS-3 was chosen because it measures adaptive behavior in a variety of domains, therefore providing a well-rounded picture of the child.

THE INTERVENTION The intervention will occur at Hearts and Horses Therapeutic Riding Center, which follows guidelines set forth by PATH, Intl to ensure safety of participants; for example, instructors are PATH-certified, trained side-walkers will be present during the intervention, and participants will wear helmets.

Prior to the intervention, each participant and caregiver will participate in an evaluation with an occupational therapist to determine current level of functioning and family priorities. Before the evaluation, caregivers will be asked to fill out two forms and bring them to the evaluation: a questionnaire about their child's adaptive functioning and the sensory profile. During the evaluation, occupational therapists will conduct a semi-structured interview with the parent and child. Next, the occupational therapist will collaborate with the child and family to create occupation-focused goals, a process that will be facilitated by the administration of the Canadian Occupational Performance Measure (COPM). Occupational therapists will help to guide the family in setting occupation-focused goals that are realistically attainable with this 10-week intervention.

Guided by the evaluation, the occupational therapist will individualize the intervention to address each participant's unique goals, accommodate for individual learning styles (e.g. minimize use of verbal cues), and incorporate each child's special interests or powerful motivators. Despite this individualization, common components will be present across all intervention sessions. Each session will be 45-60 minutes long, and the child will be mounted on the horse for at least 25 minutes. The session will begin with a visual schedule of the day's activities, which can then be referred to throughout the session to facilitate transitions from one activity to another. There will be a one-to-one ratio between the child and occupational therapist to ensure the intervention is individualized to each child's needs. Two EAOT sessions will occur simultaneously in the same arena, and the occupational therapists will facilitate social interaction between participants. Participants will be paired into groups of two so that the session that is occurring simultaneously is with a child with autism with a similar level of adaptive functioning. Activities will be structured to provide positive reinforcement for communication, and the occupational therapist will manipulate equine movement to provide graded sensory stimulation and optimal arousal. Unmounted, or "ground activities" will be customized to address each child's goal.

DATA COLLECTION: It is likely that improvements made during EAOT will be maintained after the intervention is withdrawn, therefore a multiple-baseline design is the optimal single-case experimental design. After the occupational therapy evaluation, participants will be paired into groups of two based on similar levels of adaptive functioning and/or similar or complementary treatment goals. Pairs of participants will then be randomized to a 5-week, or 7-week baseline phase. The baseline condition will be a no-treatment waiting list, during which caregivers will fill out the ABC-C on a weekly basis, retrospectively reporting on their child's behavior for the previous week. Caregivers will also complete a brief questionnaire that asks about any changes in medication, therapy, or routines that week. In addition, caregivers will rate their child's target behaviors on a VAS everyday. All of these measures (ABC-C, parent questionnaire, and VAS) will be administered online using a Qualtrics survey that is emailed or texted to them, depending on parent preference.

The 10-week intervention phase will consist of weekly, 45-minute EAOT intervention sessions. Throughout the intervention phase, caregivers will continue completing the ABC-C and brief questionnaire weekly; caregivers will also continue providing VAS ratings daily. In addition, caregivers will complete the intervention credibility scale, the SRS-2, and the COPM on the first week and the 10th week of the intervention phase, in order to provide a pre and post assessment of caregivers' attitude toward treatment, and child social functioning and occupational performance. Three months after the intervention, caregivers will complete the SRS-2, COPM, and the ABC-C a final time to determine maintenance of effects DATA ANALYSIS: Visual inspection will be the primary method of data analysis. The Co-PI will plot the dependent variables (y-axis) against time (x-axis) for each participant. Next, she will inspect the data for changes in mean (average rate of performance), and trend (direction of change over time), of the dependent variables between baseline and intervention conditions. If the data demonstrate positive findings, the plotted graphs will be further inspected for evidence of non-effect, such as delayed latency to change, positive trends during the baseline phase, or variable data with overlap between phases. As a secondary method of analysis, investigators will calculate the non-overlap of all pairs (NAP) of the ABC-C, and VAS scores between baseline and intervention phases, which will yield an effect size and a measure of statistical significance .

QUALITATIVE STRAND

PARTICIPANTS: Two occupational therapists have been recruited to participate in this study. Both occupational therapists helped to screen the children with autism to determine if they met all PATH, Intl standards for participation in equine-assisted therapy. Second, they have both helped to conduct occupational therapy evaluations to determine the current level of functioning and therapy goals for the children with autism. Third, they will provide the equine-assisted occupational therapy to children with autism. Finally, they will participate in interviews about the theory guiding the intervention they are delivering.

DATA COLLECTION & ANALYSIS: Qualitative data will consist of interviews with the occupational therapists during and after the 10-week intervention. During the course of the 10-week intervention, the Co-PI will interview both occupational therapists using a semi-structured interview guide. Overall during the intervention phase, investigators will conduct 5 hours of interviews with each occupational therapist. After the 10-week intervention has concluded and quantitative data have been analyzed, the Co-PI will conduct one final hour-long interview with both occupational therapists aimed at explaining the quantitative results.

Investigators will transcribe audio-recorded interviews and perform theoretical thematic analysis with constant comparison using the qualitative data analysis software program, NVivo. First, interviews will be coded according to these start codes, derived from work on theory-guided interventions: 1- "problems" experienced by participants 2- intervention components designed to address problems, 3- theories of change and mediational processes, and 4- intended outcomes. Next, investigators will conduct open coding, whereby the text will be broken down, examined, conceptualized, and categorized. Data will be sub-categorized within existing start-codes as appropriate, and new categories may emerge from the data. After open coding, investigators will engage in axial coding, seeking to find links and relationships between and within categories and sub-categories. Investigators will bring emerging analyses to the practitioners for occasional member checks, in order to ensure that ongoing analyses are consistent with their intended meanings. Finally, selective coding will allow final themes to emerge, and will elucidate relationships between themes.

ELIGIBILITY:
Inclusion Criteria:

* aged 5-14
* have an ASD diagnosis by a community provider
* score ≥15 on the Social Communication Questionnaire
* score ≥11 on the Aberrant Behavior Checklist-Community
* meets clinical cut-offs for ASD on the Autism Diagnostic Observation Schedule, Second Edition
* score ≥55 on the Leiter International Performance Scale, Third Edition
* can tolerate a helmet
* can participate in 10-minutes of riding while following safety rules
* meets physical, mental, and emotional standards set forth by the Professional Association of Therapeutic Horsemanship, International

Exclusion Criteria:

* behavioral issues that could interfere with safety
* 2 hours or more of previous experience with equine-assisted interventions in the last 6 months
* weight exceeding 200 pounds

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) ratings of individualized occupational performance goals | daily, during baseline and intervention phases (up to 119 days)
  Parents rate their child's performance on an individualized goal using a sliding scale. The minimum score of 0, indicated on the left of the scale, denotes poor performance, while the maximum score 100, on the right of the scale, denotes excellent performance.

SECONDARY OUTCOMES:
Change in Irritability | Weekly during baseline and intervention phases, up to 18 weeks. Also during 3-month follow-up.
  Irritability subscale of the Aberrant Behavior Checklist- Community (ABC-C). The minimum score of 0 denotes an absence of irritable behaviors, while to maximum score of 45 denotes frequent and severe irritable behaviors.
Change in Hyperactivity | Weekly during baseline and intervention phases, up to 18 weeks. Also at 3-month follow up.
  Hyperactivity subscale of the Aberrant Behavior Checklist- Community (ABC-C). The minimum score of 0 denotes an absence of hyperactive behaviors, while the maximum score of 48 denotes frequent and severe hyperactive behaviors.
Change in Social Functioning | 4 Time Points: initial, after 5-7 weeks of no-treatment baseline, after 10 weeks of intervention, and after a 3-month follow-up period.
  Parent ratings on the Social Responsiveness Scale, Second Edition. The scale ranges from 0 - 195, where higher scores indicate more social impairment.
Change in Canadian Occupational Performance Measure | 4 Time Points: initial, after 5-7 weeks of no-treatment baseline, after 10 weeks of intervention, and after a 3-month follow-up period.
  Parent ratings of performance and satisfaction with their child's progress towards individualized goals. Administered in a semi-structured interview format. Ratings range from 0 - 10, where larger scores indicate better performance or higher levels of satisfaction.

OTHER OUTCOMES:
Parent Perceptions of Child's Response to Treatment | Two time points: 1-2 months after the intervention is complete (January-February 2018) and 5 months after intervention is complete (May 2018)
  Semi-structured interviews with parents to obtain their perceptions of the therapy
Therapist Clinical Reasoning | Weekly basis for 10 weeks throughout intervention phase.
  Semi-structured interviews with therapists to understand their clinical reasoning guiding how the intervention was designed and delivered

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Wood, Ph.D., Principal Investigator — Colorado State University
Locations (1):
- Hearts and Horses Therapeutic Riding Center, Loveland, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aman MG, Singh NN, Stewart AW, Field CJ. The aberrant behavior checklist: a behavior rating scale for the assessment of treatment effects. Am J Ment Defic. 1985 Mar;89(5):485-91. PMID 3993694
- [Background] Gabriels RL, Pan Z, Dechant B, Agnew JA, Brim N, Mesibov G. Randomized Controlled Trial of Therapeutic Horseback Riding in Children and Adolescents With Autism Spectrum Disorder. J Am Acad Child Adolesc Psychiatry. 2015 Jul;54(7):541-9. doi: 10.1016/j.jaac.2015.04.007. Epub 2015 May 5. PMID 26088658
- [Background] Gotham K, Risi S, Dawson G, Tager-Flusberg H, Joseph R, Carter A, Hepburn S, McMAHON W, Rodier P, Hyman SL, Sigman M, Rogers S, Landa R, Spence MA, Osann K, Flodman P, Volkmar F, Hollander E, Buxbaum J, Pickles A, Lord C. A replication of the Autism Diagnostic Observation Schedule (ADOS) revised algorithms. J Am Acad Child Adolesc Psychiatry. 2008 Jun;47(6):642-651. doi: 10.1097/CHI.0b013e31816bffb7. PMID 18434924
- [Background] Lord, C., Rutter, M., DiLavore, P., RISI, S., Gotham, K., & Bishop, S. (2012). Autism Diagnostic Observation Schedule, Second Edition. Los Angeles, CA: Western Psychological Services.
- [Background] Roid, G. H., & Miller, L. J. (1997). Leiter International Performance Scale- Revised. Wood Dale, IL: Stoelting.
- [Background] Rutter, M., & Bailey, A. (2003). Social Communication Questionnaire. Los Angeles, CA: Western Psychological Services.
- [Background] Tsatsanis KD, Dartnall N, Cicchetti D, Sparrow SS, Klin A, Volkmar FR. Concurrent validity and classification accuracy of the Leiter and Leiter-R in low-functioning children with autism. J Autism Dev Disord. 2003 Feb;33(1):23-30. doi: 10.1023/a:1022274219808. PMID 12708577
- [Background] Kazdin, A. E. (2011). Single-case research designs: Methods for clinical and applied settings . Oxford University Press.
- [Background] Kratochwill TR, Levin JR. Enhancing the scientific credibility of single-case intervention research: randomization to the rescue. Psychol Methods. 2010 Jun;15(2):124-44. doi: 10.1037/a0017736. PMID 20515235
- [Background] Byiers BJ, Reichle J, Symons FJ. Single-subject experimental design for evidence-based practice. Am J Speech Lang Pathol. 2012 Nov;21(4):397-414. doi: 10.1044/1058-0360(2012/11-0036). Epub 2012 Oct 15. PMID 23071200
- [Background] Strauss A., & Corbin, J. (1990). Basics of Qualitative Research. Newbury Park, CA: Sage Publishing.